CLINICAL TRIAL: NCT02004171
Title: Electronic Nicotine Delivery Devices (ENDDs) or Nicotine Inhaler for Smoking Cessation
Brief Title: Electronic Cigarettes or Nicotine Inhaler for Smoking Cessation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled. Changed requirements for studying e-cigarettes.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #6863 P50DA009236-20; P50DA009236-20 (NIH)
Record Dates: First submitted 2013-11-25; First posted 2013-12-09 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2014-11

CONDITIONS: Tobacco Use Disorder
Keywords: electronic cigarette; nicotine inhaler; smoking cessation
MeSH Terms: conditions — Tobacco Use Disorder; Vaping; Smoking Cessation | interventions — Electronic Nicotine Delivery Systems; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- electronic cigarette (Experimental): electronic cigarette 24mg cartridges; 1-2 cartridges daily
  Interventions: Other: electronic cigarette
- nicotine inhaler (Active Comparator): nicotine inhaler 10mg cartridge; max 16 cartridges daily
  Interventions: Drug: nicotine inhaler

INTERVENTIONS:
Other: electronic cigarette — V2 Cigs with 24 mg nicotine cartridges
  Arms: electronic cigarette
Drug: nicotine inhaler — nicotine inhaler with 10 mg nicotine cartridges
  Other Names: Nicotrol inhaler
  Arms: nicotine inhaler

SUMMARY:
Electronic cigarettes have shown promise but have yet to proven effective for smoking cessation. This trial will evaluate the effectiveness of electronic cigarettes in smokers who are trying to quit smoking compared with a standard therapy, the nicotine inhaler. The investigators hypothesize that electronic cigarettes will be comparable to the nicotine inhaler in terms of smoking cessation.

DETAILED DESCRIPTION:
Cigarette smoking remains the leading cause of preventable death and disease worldwide.

The purpose of this trial is to evaluate the effectiveness of electronic cigarettes for smoking cessation compared to a similar nicotine replacement therapy, the nicotine inhaler.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 year old
* Meet DSM-IV criteria for nicotine dependence
* Seeking treatment for smoking cessation
* Smoking at least 15 cigarettes per day
* Capable of giving informed consent and complying with study procedures

Exclusion Criteria:

* Lifetime history of DSM-IV diagnosis of schizophrenia, schizoaffective disorder, and bipolar disorder or current diagnosis of major depressive disorder
* Current DSM-IV criteria for any other psychiatric disorder that may, according to the investigator's judgment, require either pharmacological or non- pharmacological intervention over the course of the study
* Currently receiving any treatment for nicotine dependence, including nicotine replacement therapy
* Pregnancy, lactation, or failure to use adequate contraception methods in women who are currently having sex with men
* Unstable medical condition, such as uncontrolled hypertension, angina, and oropharyngeal conditions which may make participation hazardous
* Current DSM-IV diagnosis of substance dependence, other than nicotine
* Use of cannabis or alcohol on more than 20 days in the past 30 days
* Risk for suicide

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Cigarettes smoked over 24 hours | 4 weeks

SECONDARY OUTCOMES:
Symptoms of nicotine withdrawal | 4 weeks
  We will measure the incidence and severity of nicotine withdrawal symptoms, including irritability, anxiety, depressed mood and increased appetite.
Benefits from smoking cessation | 4 weeks
  we will measure perceived benefits from smoking cessation including improved breathing, improved sense of taste and smell, and improved physical fitness.
Adverse reaction to nicotine inhaler or electronic cigarette | 4 weeks
  we will assess for any possible side effect from the electronic cigarette or the nicotine inhaler, including irritation of the mouth and throat and cough.

OTHER OUTCOMES:
Body mass index | 4 weeks
  We will measure if body mass increases as a consequence of smoking cessation.

CONTACTS AND LOCATIONS:
Overall Officials: Barney Vaughan, MD, Principal Investigator — New York State Psychiatric Institute/Columbia University
Locations (1):
- Substance Treatment and Research Services (STARS), New York, New York, United States